CLINICAL TRIAL: NCT06842628
Title: Promoting Positive Emotions and Savoring in the Elderly Through an Online Self-help Intervention: a Controlled Study.
Brief Title: Savor-Aging: the Art of Savoring Positive Emotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Daniela Villani, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 128/24
Record Dates: First submitted 2025-02-13; First posted 2025-02-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Aging Well; Positive Affect
Keywords: Savoring; Positive Aging; Positive Emotions; Positive Technology; Self-help

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Savoring Group (Experimental): Participants will complete the online savoring training for 3 weeks, by doing 2 activities per week. The exercises will be focused on savoring past, present and future time.
  Interventions: Other: Savoring
- Emotional Induction group (Active Comparator): Participants will complete six emotional induction exercises.
  Interventions: Other: Positive Emotional Induction

INTERVENTIONS:
Other: Savoring — Participants will follow an e-savoring training for 3 weeks. The first week will be focused on savoring past positive experiences (positive reminiscence and life lessons); the second week will be focused on savoring the present (absorption during an activity and writing a letter of gratitude to a significant person); and the third week will be focused on savoring the future (anticipating positive future events and making kind gestures to a significant person). After each activity, they will be guided to reflect and savor the positive emotions that emerge from the activity.
  The participants will complete some questionnaires at baseline, post-intervention, and in the one-month follow-up.
  Arms: E-Savoring Group
Other: Positive Emotional Induction — Participants will follow a positive emotional induction training for 3 weeks, with 2 exercises per week.
  The first week, they will listen to a piece of music and watch a video that elicits positive emotions; the second week, they will do an activity that they particularly enjoy in solitude and listen to a narrative about gratitude; the third week, they will listen to a narrative about hope and carry out an activity they like with a loved one. The participants will complete some questionnaires at baseline, post-intervention, and in the one-month follow-up.
  Arms: Emotional Induction group

SUMMARY:
This study is part of the larger project to promote positive aging (PNRR Age-IT Project) in the elderly through the amplification of positive experiences and emotions. This study aims to evaluate the feasibility and preliminary effects in terms of effectiveness of the "Savoring: the art of savoring positive emotions project", which is a self-help e-savoring training aimed at increasing psychological and subjective well-being in elderly participants. As secondary goals, this study aims to decrease depression and feelings of loneliness. An additional objective is to investigate user experience regarding the online protocol. A between-subjects design will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60
* Adequate understanding of the Italian language
* Possession of a technological tool to be able to access the Internet

Exclusion Criteria:

* Having a score below 26 on the MMSE that will be administered by telephone (Itel-MMSE) before division into the two groups. The Itel-MMSE scores will be converted into MMSE scores.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction With Life Scale (SWLS) | This questionnaire will be administered in T0 (baseline), T1 (post intervention - after 3 weeks) and T2 (one-month follow up).
  This scale was designed by Diener and colleagues (1985; Italian version: Di Fabio & Busoni, 2009) to investigate life satisfaction and consists of 5 items that can be answered through a 7-step Likert scale ranging from 1 "strongly disagree" to 7 "strongly agree."
Scale of Positive and Negative Experiences (SPANE) | This questionnaire will be administered in T0 (baseline), T1 (post-intervention - after 3 weeks) and T2 (one-month follow-up).
  This self-report scale consists of 12 items and was developed by Diener and colleagues (2010; Italian version: Corno, Molinari, & Baños, 2016) to measure positive and negative affect. It is composed of two sub-scales: the first refers to positive emotions (6 items: positive, good, pleasant, happy, joyful, satisfied) and the second to negative emotions (6 items: negative, bad, unpleasant, sad, fearful, angry). It can be answered through a 5-step Likert scale where 1 means "very rarely or never" and 5 means "very often or always."
Flourishing Scale (FS) | his questionnaire will be administered in stages T0 (baseline), T1 (post-intervention - after 3 weeks) and T2 (one-month follow-up)
  This scale, developed by Ryan and Deci (2001; Italian version Di Fabio, 2010), aims to investigate the elements that make up psychological well-being, including relationships, self-esteem, life purpose and optimism. It consists of 8 items and each is positively worded and responses are measured on a 7-step Likert scale, where 1 means "strongly disagree" and 7 means "strongly agree." The score range is from 8 to 56.

SECONDARY OUTCOMES:
DeJong Gierveld Loneliness Scale | This instrument will be administered in T0 (baseline), T1 (post-intervention - after 3 weeks) and T2 (one-month follow-up).
  This self-report scale, developed by Jong-Gierveld and van Tilburg (2006), assesses through 6 items social loneliness, which occurs when an individual lacks a larger social network, and emotional loneliness, caused by the lack of more intimate relationships. For each statement, the participant must express his or her degree of agreement on a 5-point Likert scale, where 0 means "Absolutely true" and 4 means "Absolutely not true" A higher score corresponds to a lower perception of social and emotional loneliness. For the purpose of this study, the items were translated into Italian from the original 6-item English version.
Center for Epidemiologic Studies- Depression Scale (CES-D) | This scale will be administered in T0 (baseline), T1 (post-intervention - after 3 weeks) and T2 (one-month follow up).
  Developed by Radloff (1977), it is a 20-item self-report scale used as a screening tool for depression in the elderly. For the purpose of this study, the 10-item short version, validated by Andersen and colleagues in 1994, will be used. Participants will be asked to indicate on a 5-step Likert scale, where 0 corresponds to "never or almost never" (less than 1 day), 1 corresponds to "sometimes or infrequently" (1-2 days), 2 corresponds to "occasionally or for a moderate amount of time" (3-4 days), and 4 corresponds to "most of the time or all of the time" (5-7 days), how they have been feeling in recent weeks. For the purpose of this study, the items have been translated into Italian.
Perceived Usefulness and Pleasantness of the Exercises | Immediately after each of the 6 activities of the training
  - Item ad hoc to investigate perceived usefulness and pleasantness of the exercise just done. After each activity of the training, participants will be asked to rate perceived usefulness and pleasantness through a 7-step Likert scale where 1 corresponds to "very little" and 7 to "very much."
User Experience | This questionnaire will be administered at T1 (post-intervention - after 3 weeks from baseline).
  A 5-item questionnaire, scored on a 7-step Likert scale, where 1 corresponds to "not at all" and 7 to "very much," will be proposed, aimed at investigating the subject's experience of using the website. In particular, the degree of aesthetic pleasantness of the website, its functionality, and the ability to engage the user will be investigated.
Perceived Usefulness of the Training | This questionnaire will be administered at T1 (post-intervention - after 3 weeks from baseline).
  The perceived usefulness of the training will be measured through a single item ("Referring to the entire training, how useful do you think it was for you?") that can be answered through a 7-step Likert scale where 1 corresponds to "very little" and 7 to "very much." In addition, there will be a section where it will be possible to express a reflection regarding the evaluation provided.
Usefulness and Pleasantness of the exercises when the training is completed | These items will be administered at T2 (one-month follow-up).
  Two items ad hoc will be administered to investigate which exercise they found most useful and which was the most enjoyable, specifying their reasons. In addition, they will be optionally asked to express a general reflection on the exercise they did. These ad hoc items will be differentiated according to their group. In fact, for the experimental group, reference will be made to the exercises proposed in the e-savoring training, while for the control group, positive emotion induction activities will be reported. The aim of these final items is to understand which exercises were found most useful and enjoyable overall by the participants, both in the control and experimental groups, so as to take them into account for future studies.
Frequency of Use of the exercises learned during the training | This item will be administred in T2 (one-month follow - up).
  Participants will be asked about the frequency with which they have put into practice in the last month the exercises experienced during the training for both the experimental and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Università Cattolica del Sacro Cuore, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villani D, Pancini E, Pesce F, Scuzzarella L. Savoring life during pandemic: an online intervention to promote well-being in emerging adults. BMC Psychol. 2023 Jul 4;11(1):196. doi: 10.1186/s40359-023-01225-z. PMID 37403128
- [Background] Salces-Cubero IM, Ramirez-Fernandez E, Ortega-Martinez AR. Strengths in older adults: differential effect of savoring, gratitude and optimism on well-being. Aging Ment Health. 2019 Aug;23(8):1017-1024. doi: 10.1080/13607863.2018.1471585. Epub 2018 May 21. PMID 29781723
- [Background] Gaggioli A, Villani D, Serino S, Banos R, Botella C. Editorial: Positive Technology: Designing E-experiences for Positive Change. Front Psychol. 2019 Jul 9;10:1571. doi: 10.3389/fpsyg.2019.01571. eCollection 2019. No abstract available. PMID 31338053
- [Background] Bryant FB, Osowski KA, Smith JL. Gratitude as a Mediator of the Effects of Savoring on Positive Adjustment to Aging. Int J Aging Hum Dev. 2021 Apr;92(3):275-300. doi: 10.1177/0091415020919999. Epub 2020 May 5. PMID 32370635